CLINICAL TRIAL: NCT00696176
Title: Preliminary Assessment of the Safety and Biological Activity of Intratumoral STAT3 DECOY in Surgically Resectable Head and Neck Squamous Cell Carcinoma
Brief Title: STAT3 DECOY in Head and Neck Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07-022
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2012-09

CONDITIONS: Head and Neck Cancer
Keywords: STAT 3 DECOY
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): STAT 3 decoy administration
  Interventions: Drug: STAT 3 DECOY

INTERVENTIONS:
Drug: STAT 3 DECOY — single administration to a head and neck tumor

SUMMARY:
The primary goal of this study is to evaluate the safety of a transcription factor decoy targeting Signal Transducer and Activator of Transcription 3(STAT3) in patients with head and neck cancer. The rationale for targeting STAT3 using this approach is to decrease STAT3-mediated gene regulation. The study has the following scientific objectives:

1. To assess the safety of a single dose of intratumoral STAT3 decoy.
2. To estimate the effect of STAT3 decoy therapy on STAT3 activation levels, STAT3-mediated gene expression, and apoptosis in treated tumors.

DETAILED DESCRIPTION:
The decision to proceed with an exploratory IND study to be conducted in a phase 0 setting was based upon the expectation that the trial will involve very limited human exposure to the STAT3 decoy, and as administered, will have no therapeutic or diagnostic intent. Rather, the trial is designed to determine if intratumoral administration of the STAT3 decoy in human head and neck tumors inhibits STAT3 target gene expression. Given the cumulative evidence supporting STAT3 as a therapeutic target in cancer, and the absence of any clinical trial to date using a STAT3 inhibitor, it was felt that there would be utility in a proof of principal study to determine if the STAT3 decoy inhibits the expression of STAT3 target genes in human head and neck cancers. To support the proposed study design, the Grandis lab carried out a kinetic study in a xenograft model of SCCHN. Preliminary results demonstrated that administration of the STAT3 decoy, but not the mutant control decoy, decreased expression of STAT3 target genes (Bcl-xL and/or Cyclin D1) at time points ranging from 1 to 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of head and neck squamous cell carcinoma(primary or recurrent) amenable to surgical resection.
* ECOG performance status of 0, 1, or 2.
* Adequate organ function
* Age greater than or equal to 18 years
* Written informed consent.
* Patients with second primary lesions will be eligible for this trial.
* Negative pregnancy test, nonlactating, and using effective means of contraception if childbearing potential.

Exclusion Criteria:

* Subjects who fail to meet the above criteria.
* Subjects who are pregnant.
* Subjects with an ECOG performance status >2.
* Subjects with tumors that are too small to biopsy prior to resection and reserve a portion of the resected specimen for research purposes.
* Subjects who receive neoadjuvant radiotherapy and/or chemotherapy within four week prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of a single injection. | pre and post surgery

SECONDARY OUTCOMES:
Evaluate the biological activity by observing the consequences of STAT3 decoy administration on STAT3 activation and target gene expression in the tumor. | pre and post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Grandis, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Sen M, Thomas SM, Kim S, Yeh JI, Ferris RL, Johnson JT, Duvvuri U, Lee J, Sahu N, Joyce S, Freilino ML, Shi H, Li C, Ly D, Rapireddy S, Etter JP, Li PK, Wang L, Chiosea S, Seethala RR, Gooding WE, Chen X, Kaminski N, Pandit K, Johnson DE, Grandis JR. First-in-human trial of a STAT3 decoy oligonucleotide in head and neck tumors: implications for cancer therapy. Cancer Discov. 2012 Aug;2(8):694-705. doi: 10.1158/2159-8290.CD-12-0191. Epub 2012 Jun 20. PMID 22719020